CLINICAL TRIAL: NCT06863987
Title: A Randomized, Multicenter, Double-Blind, Placebo-Controlled, Phase III Study to Evaluate the Efficacy and Safety of Valsartan Oral Solution in Children and Adolescent Hypertensive Patients
Brief Title: A Phase III Clinical Study of Valsartan Oral Solution for the Treatment of Hypertension in Children and Adolescents
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Shandong New Time Pharmaceutical Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NTP-XST-OS-Ⅲ
Record Dates: First submitted 2025-03-04; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — Valsartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Valsartan Oral Solution (Experimental): Screening Period: all subjects eligible for enrollment at Visit V1 received a 7-day placebo introductory period; Trial drug administration period: subjects eligible for enrollment received a half-dose of valsartan oral solution for one week after visit V2, after which subjects received a full-dose of valsartan oral solution for five weeks, with subjects required to come in for checkups at visits V3 and V4, and subjects were followed up by telephone for medication at visit V5; Randomized Placebo Withdrawal Period: two weeks of receiving valsartan oral solution after randomization at Visit V6, with telephone follow-up of subjects on medication at Visit V7 and subjects required to come to the hospital for check-ups at Visit V8; Safety observation period: after V8 visit, subjects assessed by the investigator to be able to continue the medication and who volunteered to participate in a follow-up study continued to take valsartan oral solution up to 3 months or withdrew early.
  Interventions: Drug: Valsartan Oral Solution
- Placebo (Placebo Comparator): Screening Period: all subjects eligible for enrollment at Visit V1 received a 7-day placebo introductory period; Trial drug administration period: subjects eligible for enrollment received a half-dose of valsartan oral solution for one week after visit V2, after which subjects received a full-dose of valsartan oral solution for five weeks, with subjects required to come in for checkups at visits V3 and V4, and subjects were followed up by telephone for medication at visit V5; Randomized Placebo Withdrawal Period: two weeks of receiving placebo after randomization at Visit V6, with telephone follow-up of subjects on medication at Visit V7 and subjects required to come to the hospital for check-ups at Visit V8; Safety observation period: after V8 visit, subjects assessed by the investigator to be able to continue the medication and who volunteered to participate in a follow-up study continued to take valsartan oral solution up to 3 months or withdrew early.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Valsartan Oral Solution — Valsartan oral solution, taken by mouth, once daily. It is recommended that the medication be administered at the same time each day (e.g., in the morning).
  The dose administered is based on the subject's weight at the V1 visit:
  Halve dose:
  <35 kg: 7 mL (equivalent to valsartan 20 mg);
  * 35 kg: 13 mL (equivalent to valsartan 40 mg).
  Full dose:
  <35 kg: 13 mL (equivalent to valsartan 40 mg);
  * 35 kg: 27 mL (equivalent to valsartan 80 mg).
  Arms: Valsartan Oral Solution
Drug: Placebo — placebo, taken by mouth, once daily. It is recommended that the medication be administered at the same time each day (e.g., in the morning).
  The dose administered is based on the subject's weight at the V1 visit:
  Full dose:
  <35 kg: 13 mL ;
  * 35 kg: 27 mL .
  Placebo dosing during elution phase:
  <35 kg: 7 mL;
  * 35 kg: 13 mL.
  Arms: Placebo

SUMMARY:
This study was an randomized, double-Blind, placebo-controlled, multicenter Phase II/III study.

DETAILED DESCRIPTION:
The trial was divided into three parts: a screening period, a treatment period, and an open-label safety observation period, in which the screening period consisted of screening and placebo elution, and the treatment period consisted of the test drug administration period and a randomized placebo withdrawal period.the entire trial process lasts at least 3 months (excluding the screening period).

ELIGIBILITY:
Inclusion Criteria:

1. 6 years old ≤ age ≤ 17 years old, male or female;
2. 18kg ≤ weight ≤ 160kg;
3. Initial diagnosis of essential hypertension or previous history of essential hypertension at the V1 visit, mean seated systolic blood pressure (MSSBP) and/or mean seated diastolic blood pressure (MSDBP) before the first administration of medication (at the V2 visit) at least in the 95th percentile for the same age, sex, and height (with reference to the "Chinese Guidelines for the Prevention and Control of Hypertension, Revised Edition 2018" for Chinese children aged 3-17 years for each year of age, height corresponding blood pressure standard) and meets the criteria for hypertension medication;
4. Vital organ function meets the following requirements:

   Blood routine: hemoglobin ≥ 90 g/L, platelet count ≥ 100 × 109 /L, serum potassium ≤ 5.3 mmol/L; Liver function: ALT and AST ≤ 3 × ULN, total bilirubin level (TBIL) ≤ 2 × ULN; Renal function: glomerular filtration rate ≥ 30 mL/min/1.73 m2 (see Appendix 1 for calculation formula);
5. The legal guardian and/or the person himself/herself voluntarily signed the informed consent form.

Exclusion Criteria:

1. those with confirmed or previous hypertensive emergencies, hypertensive sub-emergencies;
2. Patients with secondary hypertension;
3. Medication adherence <80% and/or >120% during the placebo washout period at the V2 visit;
4. Patients with diabetes mellitus judged uncontrollable by the investigator;
5. Persons with associated electrolyte disturbances (e.g., severe hyponatremia);
6. those with a prior history of biliary cirrhosis and cholestasis;
7. persons with a prior history of organ transplantation;
8. patients with known active gastritis, duodenal ulcer or gastric ulcer or gastrointestinal/rectal bleeding within 3 months prior to the first dose;
9. Patients with a history of clinically significant drug/food allergy (within 6 months prior to first dose) or history of atopic allergic disease (e.g., asthma, etc.) or known allergy to valsartan and its excipients or other angiotensin II receptor antagonists (ARBs) and/or angiotensin converting enzyme inhibitors (ACEIs);
10. Persons who are infectious disease screen positive for hepatitis B surface antigen and/or core antibody and test positive for HBV-DNA, hepatitis C virus antibody positive and test positive for RNA, HIV positive, or syphilis spirochete antibody positive;
11. Persons who have been treated with any other clinical trial drug/device within 1 month prior to the first dose or within 5 half-lives of the trial drug, whichever is shorter;
12. Females with a history of menstruation who have had a positive pregnancy test;
13. Those who may not be able to complete the study for other reasons or those who, in the opinion of the investigator, are not suitable for inclusion.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 342 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in mean seated systolic blood pressure (MSSBP) from the end of week 6 to the end of week 8 in the valsartan oral solution group compared to the placebo group. | 2 weeks of randomized placebo withdrawal period

SECONDARY OUTCOMES:
Change in mean seated diastolic blood pressure (MSDBP) from the end of week 6 to the end of week 8 | 2 weeks of randomized placebo withdrawal
Change in MSSBP and MSDBP from baseline to the end of week 6 | 6 weeks of Trial drug administration period
Change in MSSBP and MSDBP from baseline to the end of week 8 | 8 weeks of Trial drug administration period and randomized placebo withdrawal period
Blood pressure control rate | 8 weeks of Trial drug administration period and randomized placebo withdrawal period
Adverse events (AEs)/serious adverse events (SAEs) were collected by vital signs, physical examination, laboratory tests, and 12-lead electrocardiogram to assess safety | up to 3 months
Palatability evaluation by VAS (visual analog scale) | the first 8 days of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong New Time Pharmaceutical Co.LTD,, Linyi, Shandong, China

IPD SHARING:
Plan to Share IPD: No